CLINICAL TRIAL: NCT00326313
Title: Clinical Outcome of Neonate With GBS Positive Culture-12 Year Retrospective Study
Brief Title: Clinical Outcome of Neonates With GBS Positive Culture-12 Year Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4132-TS-CTIL
Record Dates: First submitted 2006-05-14; First posted 2006-05-16 (Estimated); Last update posted 2006-05-16 (Estimated); Status verified 2006-05

CONDITIONS: Infants With Positive GBS Bacteremia
Keywords: Group B streptococci; virulent; morbidity; mortality

SUMMARY:
Streptococci group B (GBS) is a the major reason for morbidity and mortality in neonates. It can present as pneumonia ,meningitis or sepsis.The mortality today is 5-20% and even more in preterm babies.

During the past two decade, the introduction of protocols for prophylactic antibiotics for women with a high risk for GBS infection, have led to a decline of 65% in GBS cases(0.32 for 1000 live birth compared to 1.8 cases in 1000).The purpose of the study is to check the morbidity and mortality at Sheba medical center in the last 12 years in children with positive blood culture for GBS. We assume that in our hospital the morbidity and mortality is less then expected. If proven right, we would then check the reasons for that outcome considering the type and length of treatment and the different virulence of the streptococcus.

DETAILED DESCRIPTION:
This is a retrospective case control study. We will review from archive the charts of all the neonates with positive blood culture for GBS, reviewing the course and severity of their illness.

ELIGIBILITY:
Inclusion Criteria:

* GBS positive blood culture neonate and preterm babies

Exclusion Criteria:

* Congenital malformations

Ages: 0 Years to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Tzipora Strauss, MD, Principal Investigator — Sheba Medical Center